CLINICAL TRIAL: NCT04936607
Title: ImproviNg rEnal Outcomes Following Coronary angiograPhy and/or percuTaneoUs coroNary intErventions: a Pragmatic, Adaptive, Patient-oriented Randomized Controlled Trial
Brief Title: ImproviNg rEnal Outcomes Following Coronary angiograPhy and/or percuTaneoUs coroNary intErventions
Acronym: NEPTUNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Université de Montréal (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Guillaume Marquis-Gravel, Assistant professor, Université de Montreal, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ICM 2022-2949
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Contrast-Induced Acute Kidney Injury
Keywords: Randomized controlled trial; Pragmatic trial; Adaptive trial; Patient-oriented trial; Contrast-induced Nephropathy; Acute Kidney Injury; Coronary angiography; Percutaneous coronary intervention
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personnalized hydration strategy (Experimental): In the experimental group, NS infusion rate will be adjusted based on LVEDP for the whole duration of the procedure (<13 mmHg: 5 ml/kg/h; 13-18 mmHg: 3 ml/kg/h; >18 mmHg: 1.5 ml/kg/h), or for one hour, whichever is the longest. After the procedure, and for a duration of 4 hours, the hydration rate will be adjusted based on the (contrast volume:estimated glomerular filtration rate (eGFR)) ratio, according to the following scheme: 1.5 ml/kg/h if contrast volume/eGFR ratio <2.0; 3 ml/kg/h for contrast volume/eGFR ratio 2.0-2.9; 5 ml/kg/h for contrast volume/eGFR ratio ≥3.0.
  Interventions: Procedure: Personalized hydration strategy
- Standard of care (Active Comparator): In the control group, infusion rate will be of 1.5 ml/kg/h during the procedure, and for the 4 following hours.
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Procedure: Personalized hydration strategy — In the experimental group, NS infusion rate will be adjusted based on LVEDP for the whole duration of the procedure (<13 mmHg: 5 ml/kg/h; 13-18 mmHg: 3 ml/kg/h; >18 mmHg: 1.5 ml/kg/h), or for one hour, whichever is the longest. After the procedure, and for a duration of 4 hours, the hydration rate will be adjusted based on the (contrast volume:estimated glomerular filtration rate (eGFR)) ratio, according to the following scheme: 1.5 ml/kg/h if contrast volume/eGFR ratio <2.0; 3 ml/kg/h for contrast volume/eGFR ratio 2.0-2.9; 5 ml/kg/h for contrast volume/eGFR ratio ≥3.0.
  Arms: Personnalized hydration strategy
Procedure: Standard of care — In the control group, infusion rate will be of 1.5 ml/kg/h during the procedure, and for the 4 following hours.
  Arms: Standard of care

SUMMARY:
The NEPTUNE triple-blind, active-placebo, adaptive, pragmatic, randomized trial aims to evaluate the effectiveness of a new intra-venous hydration strategy guided by left ventricular end-diastolic pressure (LVEDP), amount of contrast used, and baseline renal function, to prevent contrast-induced acute kidney injury (CI-AKI) and patient-oriented clinical endpoints in all-comer patients undergoing coronary angiogram and/or percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
All-comer patients undergoing a coronary angiogram and/or a PCI and meeting the eligibility criteria will be randomized to be treated with either a hydration strategy personalized to LVEDP, amount of contrast used, and baseline renal function, or to standard, non-tailored hydration (1:1 allocation ratio stratified by GFR ≥60 vs. <60 mL/min/1.73 m2). The operators (interventional cardiologists and fellows) and the participants will be blinded to the treatment allocation during the procedure. Serum creatinine will be measured at 48 hours, 7 days, and 6 months after the procedure, and the incidence of contrast-induced acute kidney injury (CI-AKI) (primary endpoint) and of major adverse renal and cardiovascular events will be evaluated by a blinded and independent expert adjudication committee.

All participants will be treated with a commercially available 0.9% NaCl solution (normal saline, NS) infusion at a rate of 3 mL/kg/h for one hour prior to the procedure. In both study groups, LVEDP will be measured at the beginning of the procedure by introducing a catheter in the left ventricle, as performed routinely in clinical practice. In the experimental group, NS infusion rate will be adjusted based on LVEDP for the whole duration of the procedure (<13 mmHg: 5 ml/kg/h; 13-18 mmHg: 3 ml/kg/h; >18 mmHg: 1.5 ml/kg/h), or for one hour, whichever is the longest. After the procedure, and for a duration of 4 hours, the hydration rate will be adjusted based on the (contrast volume:estimated glomerular filtration rate (eGFR)) ratio, according to the following scheme: 1.5 ml/kg/h if contrast volume/eGFR ratio <2.0; 3 ml/kg/h for contrast volume/eGFR ratio 2.0-2.9; 5 ml/kg/h for contrast volume/eGFR ratio ≥3.0. In the control group, infusion rate will be of 1.5 ml/kg/h during the procedure, and for the 4 following hours.

This study will follow an adaptive design in which the primary endpoint will be shifted to a more patient-oriented endpoint at the time of a single interim analysis according to pre-specified criteria established in the protocol. The adaptive design will allow to stop the trial if the experimental strategy is futile to reduce the rates of CI-AKI, and to continue on an operationally seamless manner if the experimental strategy is beneficial to reduce CI-AKI, transitioning to major adverse renal and cardiovascular endpoints (MARCE) as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Planned coronary angiogram and/or PCI;
* Willingness to participate and to attend study visits;
* Expected life expectancy ≥6 months.

Exclusion Criteria:

* Cardiogenic or non-cardiogenic shock at the time of the procedure;
* Emergent procedures (e.g. STEMI);
* Iodine-based contrast media received within 2 days;
* Presence of Intra-Aortic Balloon Pump (IABP);
* Cardiac arrest within 24 hours;
* Pre-procedural AKI defined using the modified KDIGO criteria within 7 days;
* Renal replacement therapy;
* Severe aortic or mitral disease;
* LVEF <30%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1158 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Contrast-induced acute kidney injury | 7 days
  Increase in creatinine of 1.5 times baseline within 7 days or increase in creatinine by 26.5 umol/L (i.e. 0.3 mg/dL) within 48 hours

SECONDARY OUTCOMES:
Major adverse renal and cardiovascular events (MARCE) | 6 months
  Composite of death, myocardial infarction, stroke, or renal replacement therapy
MARCE composite with the addition of persistent increase of at least 50% from baseline serum creatinine | 6 months
  MARCE composite with the addition of persistent increase of at least 50% from baseline serum creatinine
All-cause death | 6 months
  All-cause death
Myocardial infarction | 6 months
  Myocardial infarction (types 1-5)
Stroke | 6 months
  Ischemic, hemorrhagic, or undetermined stroke
Renal replacement therapy | 6 months
  Any type of renal replacement therapy (dialysis, hemofiltration, hemodiafiltration, or other)
Chronic kidney disease | 6 months
  50% increase from baseline serum creatinine
Worsening of kidney disease | 6 months
  Transition to a higher KDIGO CKD stage
Hospital length-of-stay | 6 months
  Hospital length-of-stay after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Marquis-Gravel, MD, MSc, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan.